CLINICAL TRIAL: NCT03617549
Title: A Pilot Test to Evaluate the Effect of Maternal Stress on Breastmilk Quantity and Stress Biomarkers in Mothers and Their Infants
Brief Title: Stress and Breast Milk Study In the Neonatal Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Casey Rosen-Carole, Assistant Professor, University of Rochester
Other Study IDs: RSRB#000000
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Breast Feeding; Breast Milk Expression; Stress
Keywords: neonatal intensive care
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, saliva, breastmilk
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Mothers of singleton moderate preterm appropriate for Gestational Age (AGA) infants (29-32+6 weeks gestation in the neonatal intensive care unit at the Golisano Children's Hospital

SUMMARY:
The overall goal of this research is to clarify the relationship between reported maternal stress, biological measures of maternal stress, breast milk biomarkers and milk quantity. Our primary hypothesis is that measures of maternal stress are associated with cortisol, cytokines, and other stress markers in the blood, which impacts breast milk quantity and composition and which may impact infant health.

ELIGIBILITY:
Inclusion Criteria:

* Baby will remain in mom's legal custody
* Intends to exclusively breastfeed during the NICU stay
* Has kept a daily log of milk expression (pump or hand expression) with date/time/quantity since birth of their child
* Less than 7 days postpartum

Exclusion Criteria:

* Baby and mother are to be separated due to legal custody issues
* Medical contraindication to breastfeeding
* Non-English speaking
* Unable to answer a written survey in English
* More than 50% of infant intake is not mother's own milk at 4 weeks postpartum

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Mothers of singleton moderate preterm appropriate for Gestational Age (AGA) infants (29-32+6 weeks gestation29) will be approached during the enrollment period and screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Correlation between secretory IgA levels in mother's serum and reported stress | baseline
  Mother's stress will be measured using the The Parent Stress Scale: Neonatal Intensive Care Unit. This scale ranges from 1-130 with higher numbers indicating more stress.
  Serum will be collected from mothers at enrollment and 4 weeks postpartum. Maternal venipuncture will be used to collect an 0.5mL aliquot of whole blood at the time of mother's first morning pump session in the neonatal intensive care unit. IgA will be quantitated using the Millipore Magpix 100 System. Multivariate regression analysis will be used to test for correlations.
Correlation between secretory IgA levels in mother's serum and reported stress | 1 month
  Mother's stress will be measured using the The Parent Stress Scale: Neonatal Intensive Care Unit. This scale ranges from 1-130 with higher numbers indicating more stress.
  Serum will be collected from mothers at enrollment and 4 weeks postpartum. Maternal venipuncture will be used to collect an 0.5mL aliquot of whole blood at the time of mother's first morning pump session in the neonatal intensive care unit. IgA will be quantitated using the Millipore Magpix 100 System. Multivariate regression analysis will be used to test for correlations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center NICU, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No